CLINICAL TRIAL: NCT00294684
Title: A Randomized, Double-Blinded, Placebo-Controlled Trial of Corticosteroid Therapy Following Portoenterostomy in Infants With Biliary Atresia
Brief Title: A Randomized, Double-Blinded, Placebo-Controlled Trial of Corticosteroid Therapy Following Portoenterostomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CHILDREN (START) (IND); U01DK062456 (NIH)
Record Dates: First submitted 2006-02-21; First posted 2006-02-22 (Estimated); Results first posted 2017-05-05 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Biliary Atresia
Keywords: biliary atresia; hepatoportoenterostomy; corticosteroids
MeSH Terms: conditions — Biliary Atresia | interventions — Adrenal Cortex Hormones; Methylprednisolone; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Corticosteroids (Experimental)
  Interventions: Drug: Corticosteroids
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Corticosteroids — Schedule and dosing of corticosteroids following portoenterostomy in infants with biliary atresia are listed below.
  Days 1-3: Methylprednisolone, IV-4mg/kg/day, divided BID Days 4-7: Prednisolone, PO-4mg/kg/day, divided BID Week 2: 4 mg/kg/day, divided BID Week 3: 2 mg/kg/day, divided BID Week 4: 2 mg/kg/day, divided BID Week 5: 1 mg/kg/day, once a day Week 6: 1 mg/kg/day, once a day Week 7: 0.8 mg/kg/day, once a day Week 8: 0.6 mg/kg/day, once a day Week 9: 0.4 mg/kg/day, once a day Week 10: 0.2 mg/kg/day, once a day Week 11: 0.1 mg/kg/day, once a day Week 12-13: 0.1 mg/kg/day, every other day Week 14: Stop
  Other Names: methylprednisolone; prednisolone
  Arms: Corticosteroids
Drug: Placebo — Schedule and dosing of placebo following portoenterostomy in infants with biliary atresia:
  Days 1-3: IV - normal saline 4 mg/kg/day, divided BID Days 4-7: PO placebo 4 mg/kg/day, divided BID Week 2: PO placebo 4 mg/kg/day, divided BID Week 3: PO placebo 2 mg/kg/day, divided BID Week 4: PO placebo 2 mg/kg/day, divided BID Week 5: PO placebo 1 mg/kg/day, once a day Week 6: PO placebo 1 mg/kg/day, once a day Week 7: PO placebo 0.8 mg/kg/day, once a day Week 8: PO placebo 0.6 mg/kg/day, once a day Week 9: PO placebo 0.4 mg/kg/day, once a day Week 10: PO placebo 0.2 mg/kg/day, once a day Week 11: PO placebo 0.1 mg/kg/day, once a day Week 12-13: PO placebo 0.1 mg/kg/day, once a day every other day Week 14: Stop
  Arms: Placebo

SUMMARY:
The Children Liver Disease Research and Education Network (ChiLDREN) is conducting a clinical trial to evaluate whether long-term treatment with corticosteroids improves the outcome of the Kasai or gall-bladder Kasai in infants with biliary atresia. In this clinical trial, ChiLDREN is testing whether corticosteroid therapy following the Kasai will improve bile drainage and long term outcome in infants with biliary atresia. Subjects in this trial must start treatment within 72 hours of the Kasai procedure and be part of a prospective study of the natural history of biliary atresia also being conducted by ChiLDREN (http://www.clinicaltrials.gov/ct/show/NCT00061828?order=3).

DETAILED DESCRIPTION:
This is a multi-center randomized, double-blinded, placebo-controlled trial to prospectively determine the efficacy of corticosteroids on the outcome of infants with biliary atresia. The trial will be conducted by the NIDDK-funded network of 15 clinical centers comprising the Biliary Children Liver Disease Research and Education Network (ChiLDREN), whose goal is to study the etiology, pathogenesis, diagnosis, and treatment of infants with biliary atresia. For the trial, our overall hypothesis is that therapy with corticosteroids following portoenterostomy (including gall bladder Kasai procedure) will improve bile drainage and long-term outcome in infants with biliary atresia. This hypothesis will be tested through the following specific aims and hypotheses:

Aim 1: To determine whether corticosteroid therapy decreases serum bilirubin concentration after portoenterostomy.

Aim 2: To determine whether corticosteroid treatment after portoenterostomy will improve outcome as defined by survival without transplantation at 24 months of age.

Aim 3: To determine whether corticosteroid treatment after portoenterostomy will improve growth of infants with biliary atresia.

Aim 4: To determine whether corticosteroid treatment improves biochemical indicators of each of the fat-soluble vitamins after supplementation with standard doses.

Aim 5: To determine whether corticosteroid treatment after portoenterostomy will decrease the incidence of persistent ascites or ascites that requires medical treatment.

The significance of the proposed trial is that it will determine whether corticosteroids are an effective medical treatment to improve bile drainage and long-term outcome, and whether its use reduces the need for liver transplantation in infants with biliary atresia.

Subjects will be recruited from patients enrolled in the ChiLDREN prospective observational database study who undergo portoenterostomy or portochelecystostomy (gall bladder Kasai) for biliary atresia.

The Primary outcome measure is the percentage of patients with serum total bilirubin <1.5 mg/dL and with native liver at 6 months after portoenterostomy.

Secondary outcome measures are:

1. Serum total bilirubin concentration (and also at 3 months after portoenterostomy)
2. Survival with native liver at 24 months of age
3. Growth

   1. Weight for age Z-score (in patients without ascites)
   2. Height for age Z score
4. Serum biomarkers of sufficiency of fat-soluble vitamins

   1. Vitamin A: molar ratio of serum retinol/retinol binding protein
   2. Vitamin D: serum level of 25-hydroxy vitamin D
   3. Vitamin E: ratio of serum vitamin E/total lipids
   4. Vitamin K: International Normalized Ratio (INR)
5. Presence of ascites

All measurements will be made at 12 and 24 months of age (unless noted otherwise):

ELIGIBILITY:
Inclusion Criteria:

* Portoenterostomy or gall bladder Kasai operation for biliary atresia within the previous 72 hours
* Post-conception age ≥ 36 weeks
* Weight at enrolment ≥ 2000 gm
* Written informed consent to participate in the study obtained prior to or within 72 hours of completion of portoenterostomy. (Note: Families of potential subjects may be approached prior to the portoenterostomy.)

Exclusion Criteria:

* Known immunodeficiency
* Diabetes mellitus
* Presence of significant systemic hypertension for age (persistent systolic blood pressure ≥112 mmHg)
* A serum indirect (unconjugated) bilirubin ≥ 5 mg/dL for infants under 4 weeks of age or ≥ 7 mg/dL for infants between 4 and 8 weeks of age
* Known sensitivity to corticosteroids
* Documented bacteremia or other tissue infection which is felt to be clinically relevant
* Known congenital infection or disease with herpes simplex virus, toxoplasmosis, or cytomegalovirus inclusion disease of the liver
* Infants whose mother is known to have human immunodeficiency virus infection
* Infants whose mother is known to be HBsAg or hepatitis C virus positive
* Infants with other severe concurrent illnesses such as neurological, cardiovascular, pulmonary, metabolic, endocrine, and renal disorders that would interfere with the conduct and results of the study
* Any other clinical condition that is a contraindication to the use of corticosteroid (e.g., bowel perforation)
* Infants who have received the live attenuated rotavirus vaccine (e.g., Rotateq) within 5 days prior to proposed administration of study drug

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 141 (Actual)
Dates: Start 2005-11; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Sokol, MD, Study Chair — Children's Hospital Colorado; Ed Doo, MD, Study Director — National Institute of Diabetes and Digestive and Kidney Disease (NIDDK); John Magee, MD, Principal Investigator — University of Michigan Medical Center, Ann Arbor; Averell Sherker, MD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (14):
- United States (14):
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California at San Francisco, San Francisco, California
  - The Children's Hospital, Aurora, Colorado
  - Children's Hospital of Atlanta - Emory University, Atlanta, Georgia
  - Children's Memorial Hospital, Chicago, Illinois
  - Riley Children's Hospital, Indianapolis, Indiana
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Mount Sinai Medical Center, New York, New York
  - Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital at Pittsburgh, Pittsburgh, Pennsylvania
  - Texas Children's Hospital/Baylor College of Medicine, Houston, Texas
  - Children's Hospital and Regional Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Archived dataset will be entered into NIDDK Repository
Supporting Information: Study Protocol, Analytic Code
Time Frame: Within six months of the publication date for the primary outcome publication or within two years of the date that the database is locked for analysis, whichever occurs first.
URL: https://repository.niddk.nih.gov/studies/start/?query=start

REFERENCES:
- [Result] Bezerra JA, Spino C, Magee JC, Shneider BL, Rosenthal P, Wang KS, Erlichman J, Haber B, Hertel PM, Karpen SJ, Kerkar N, Loomes KM, Molleston JP, Murray KF, Romero R, Schwarz KB, Shepherd R, Suchy FJ, Turmelle YP, Whitington PF, Moore J, Sherker AH, Robuck PR, Sokol RJ; Childhood Liver Disease Research and Education Network (ChiLDREN). Use of corticosteroids after hepatoportoenterostomy for bile drainage in infants with biliary atresia: the START randomized clinical trial. JAMA. 2014 May 7;311(17):1750-9. doi: 10.1001/jama.2014.2623. PMID 24794368
- [Derived] Alonso EM, Ye W, Hawthorne K, Venkat V, Loomes KM, Mack CL, Hertel PM, Karpen SJ, Kerkar N, Molleston JP, Murray KF, Romero R, Rosenthal P, Schwarz KB, Shneider BL, Suchy FJ, Turmelle YP, Wang KS, Sherker AH, Sokol RJ, Bezerra JA, Magee JC; ChiLDReN Network. Impact of Steroid Therapy on Early Growth in Infants with Biliary Atresia: The Multicenter Steroids in Biliary Atresia Randomized Trial. J Pediatr. 2018 Nov;202:179-185.e4. doi: 10.1016/j.jpeds.2018.07.002. Epub 2018 Sep 21. PMID 30244988
- [Derived] Ng VL, Sorensen LG, Alonso EM, Fredericks EM, Ye W, Moore J, Karpen SJ, Shneider BL, Molleston JP, Bezerra JA, Murray KF, Loomes KM, Rosenthal P, Squires RH, Wang K, Arnon R, Schwarz KB, Turmelle YP, Haber BH, Sherker AH, Magee JC, Sokol RJ; Childhood Liver Disease Research Network (ChiLDReN). Neurodevelopmental Outcome of Young Children with Biliary Atresia and Native Liver: Results from the ChiLDReN Study. J Pediatr. 2018 May;196:139-147.e3. doi: 10.1016/j.jpeds.2017.12.048. Epub 2018 Mar 5. PMID 29519540
- [Derived] Shneider BL, Magee JC, Karpen SJ, Rand EB, Narkewicz MR, Bass LM, Schwarz K, Whitington PF, Bezerra JA, Kerkar N, Haber B, Rosenthal P, Turmelle YP, Molleston JP, Murray KF, Ng VL, Wang KS, Romero R, Squires RH, Arnon R, Sherker AH, Moore J, Ye W, Sokol RJ; Childhood Liver Disease Research Network (ChiLDReN). Total Serum Bilirubin within 3 Months of Hepatoportoenterostomy Predicts Short-Term Outcomes in Biliary Atresia. J Pediatr. 2016 Mar;170:211-7.e1-2. doi: 10.1016/j.jpeds.2015.11.058. Epub 2015 Dec 24. PMID 26725209
- [Derived] Venkat VL, Shneider BL, Magee JC, Turmelle Y, Arnon R, Bezerra JA, Hertel PM, Karpen SJ, Kerkar N, Loomes KM, Molleston J, Murray KF, Ng VL, Raghunathan T, Rosenthal P, Schwartz K, Sherker AH, Sokol RJ, Teckman J, Wang K, Whitington PF, Heubi JE; Childhood Liver Disease Research and Education Network. Total serum bilirubin predicts fat-soluble vitamin deficiency better than serum bile acids in infants with biliary atresia. J Pediatr Gastroenterol Nutr. 2014 Dec;59(6):702-7. doi: 10.1097/MPG.0000000000000547. PMID 25419594
- [Derived] Shneider BL, Magee JC, Bezerra JA, Haber B, Karpen SJ, Raghunathan T, Rosenthal P, Schwarz K, Suchy FJ, Kerkar N, Turmelle Y, Whitington PF, Robuck PR, Sokol RJ; Childhood Liver Disease Research Education Network (ChiLDREN). Efficacy of fat-soluble vitamin supplementation in infants with biliary atresia. Pediatrics. 2012 Sep;130(3):e607-14. doi: 10.1542/peds.2011-1423. Epub 2012 Aug 13. PMID 22891232
- See also: Children Liver Disease Research and Education Network (ChiLDREN) — http://www.childrennetwork.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One patient was enrolled but not randomized. Therefore, the overall number enrolled is 141, while the number randomized and starting participant flow is 140.
Period: Overall Study
Arm/Group | Corticosteroids | Placebo
Started | 70 | 70
Completed | 65 | 62
Not Completed | 5 | 8
Not completed — Lost to Follow-up | 5 | 8

BASELINE CHARACTERISTICS:
Population: Intent to Treat
Groups:
- Total: Total of all reporting groups
Arm/Group | Corticosteroids | Placebo | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Continuous [Mean (Standard Deviation); unit: Months] | 2.3 (.93) | 2.3 (.84) | 2.3 (.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 40 | 72
  Male | 38 | 30 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 22 | 36
  Not Hispanic or Latino | 55 | 48 | 103
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 11 | 19
  White | 46 | 44 | 90
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 16 | 15 | 31
Biliary atresia splenic malformation (BASM) [Number; unit: participants] — BASM (Biliary Atresia Splenic Malformation) categorization as provided by the study sites (absent or present). Patients where BASM is considered present are provided as "Number" below. Other patients are considered absent of BASM.
  participants
    BASM | 2 | 3 | 5
    Not BASM | 68 | 67 | 135
OHI Main Type [Number; unit: participants] — Ohi classifications are provided by the study sites. Type I = atresia of common bile duct, Type II = atresia of hepatic duct and Type III = atresia of porta hepatis.
  participants
    I | 5 | 8 | 13
    II | 1 | 4 | 5
    III | 64 | 57 | 121
    Missing | 0 | 1 | 1
Total Bilirubin [Mean (Standard Deviation); unit: mg/dL] | 7.5 (2.6) | 7.9 (2.8) | 7.7 (2.7)
Length Z Score [Mean (Standard Deviation); unit: Z-Score] | -0.7 (1.35) | -0.6 (1.35) | -0.65 (1.35)
Weight Z Score [Mean (Standard Deviation); unit: Z-Score] | -0.8 (1.07) | -0.8 (1.06) | -0.8 (1.07)

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients With Serum Total Bilirubin <1.5 mg/dL and With Native Liver at 6 Months After Portoenterostomy
Time Frame: Measurements will be made at 6 months after portoenterostomy
Population: Intent to Treat
Measure: Number; unit: percentage of participants
Arm/Group | Corticosteroids | Placebo
Number analyzed (Participants) | 70 | 70
percentage of participants | 58.6 | 48.6
Statistical Analysis 1: Comparison: Corticosteroids vs Placebo; RR greater than one indicates benefit of steriods and a P value of treatment success from a log-binomial model with these covariates: Treatment group, age a HPE, BASM as fixed effects, and site as a random effect; Test type: Superiority or Other; p = 0.43, Log binomial; Risk Ratio (RR) = 1.14, 95% CI 2-sided [0.83 to 1.57]

2. Secondary Outcome: Survival With Native Liver at 24 Months of Age
Time Frame: Measurements will be made at 24 months of age
Population: Intent to Treat
Measure: Number; unit: percentage of participants
Arm/Group | Corticosteroids | Placebo
Number analyzed (Participants) | 70 | 70
percentage of participants | 58.7 | 59.4
Statistical Analysis 1: Comparison: Corticosteroids vs Placebo; Test type: Superiority or Other; p = 0.99, Regression, Cox; Hazard Ratio (HR) = 1.0, 95% CI 2-sided [0.6 to 1.8]

3. Secondary Outcome: Serum Total Bilirubin Concentration
Time Frame: Measurements will be made at 3 months after portoenterostomy
Population: Intent to treat patients with 3 month bilirubin available are analyzed. There are no imputations for unobserved data. Patients with missing data are simply not included.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Corticosteroids | Placebo
Number analyzed (Participants) | 63 | 65
mg/dL | 3.5 (5.32) | 5.1 (6.15)
Statistical Analysis 1: Comparison: Corticosteroids vs Placebo; LS Mean difference reported as steroid minus placebo (negative values mean larger average values of total bilirubin in placebo); Test type: Superiority or Other; p = 0.0973, Mixed Models Analysis; Mean Difference (Net) = -1.6, 95% CI 2-sided [-3.49 to 0.3]

4. Secondary Outcome: Total Bilirubin Concentration at 12 Months
Time Frame: 12 Months post HPE
Population: Intent to treat patients with 12 month bilirubin available are analyzed. There are no imputations for unobserved data. Patients with missing data are simply not included.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Corticosteroids | Placebo
Number analyzed (Participants) | 41 | 36
mg/dL | 1.7 (3.63) | 3.7 (6.63)
Statistical Analysis 1: Comparison: Corticosteroids vs Placebo; LS Mean difference of steroid minus placebo (negative values indicate larger average values of bilirubin in placebo); Test type: Superiority or Other; p = 0.0552, Mixed Models Analysis; Mean Difference (Net) = -2.3, 95% CI 2-sided [-4.65 to 0.05]

5. Secondary Outcome: Total Bilirubin Concentration at 24 Months of Age
Time Frame: At 24 Months of Age
Population: Intent to treat patients with 24 month bilirubin available are analyzed. There are no imputations for unobserved data. Patients with missing data are simply not included.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Corticosteroids | Placebo
Number analyzed (Participants) | 35 | 30
mg/dL | 1.3 (3.37) | 1.6 (3.73)
Statistical Analysis 1: Comparison: Corticosteroids vs Placebo; LS Mean difference of steroid minus placebo (negative values indicate larger average bilirubin in placebo); Test type: Superiority or Other; p = 0.6607, Mixed Models Analysis; Mean Difference (Net) = -0.39, 95% CI [-2.16 to 1.38]

6. Secondary Outcome: Weight Z-Score
Description: weight for age Z-score (in subjects without ascites) over the course of the study
Time Frame: HPE until 24 months of age
Measure: Mean (Standard Error); unit: Z-score
Arm/Group | Corticosteroids | Placebo
Number analyzed (Participants) | 70 | 70
Z-score | -0.8 (0.13) | -0.8 (0.13)
Statistical Analysis 1: Comparison: Corticosteroids vs Placebo; Test type: Superiority or Other; p = 0.1603, Mixed Models Analysis

7. Secondary Outcome: Height Z-Score
Description: Height by Age Z-score over the course of the study
Time Frame: HPE to age 24 Months
Measure: Mean (Standard Error); unit: Z-score
Arm/Group | Corticosteroids | Placebo
Number analyzed (Participants) | 70 | 70
Z-score | -0.7 (0.16) | -0.6 (0.16)
Statistical Analysis 1: Comparison: Corticosteroids vs Placebo; Test type: Superiority or Other; p = 0.2801, Mixed Models Analysis

8. Secondary Outcome: Presence of Ascites at 12 Months
Time Frame: 12 Months
Population: Participants with their native liver at 12 months
Measure: Number; unit: participants
Arm/Group | Corticosteroids | Placebo
Number analyzed (Participants) | 52 | 47
participants | 5 | 3
Statistical Analysis 1: Comparison: Corticosteroids vs Placebo; Test type: Superiority or Other; p = 0.41, Log Binomial; Risk Ratio (RR) = 1.4, 95% CI 2-sided [0.62 to 3.14]

9. Secondary Outcome: Presence of Ascites at 24 Months
Time Frame: 24 Months
Population: Participants with their native liver at 24 months
Measure: Number; unit: participants
Arm/Group | Corticosteroids | Placebo
Number analyzed (Participants) | 42 | 43
participants | 1 | 3
Statistical Analysis 1: Comparison: Corticosteroids vs Placebo; Test type: Superiority or Other; p = 0.29, Log Binomial; Risk Ratio (RR) = 0.3, 95% CI 2-sided [0.03 to 2.92]

10. Other Pre Specified Outcome: Serum Biomarkers of Sufficiency of Fat-soluble Vitamins - Vitamin E
Description: Vitamin E sufficiency is measured as the ratio of serum vitamin E/total lipids
Time Frame: 24 Months
Population: Although the protocol specified analyses of serum biomarkers as secondary outcomes, the intent was to only perform these analyses if the primary endpoint showed sufficient efficacy. Given the lack of efficacy of steroids (vs placebo), the analyses of fat-soluble vitamins were not performed; thus, data are not summarized for this assessment.
Arm/Group | Corticosteroids | Placebo
Number analyzed (Participants) | 0 | 0

11. Other Pre Specified Outcome: Serum Biomarkers of Sufficiency of Fat-soluble Vitamins - Vitamin K
Description: Vitamin K sufficiency is measured by INR (international normalized ratio)
Time Frame: 24 Months
Population: as for outcome 10
Arm/Group | Corticosteroids | Placebo
Number analyzed (Participants) | 0 | 0

12. Other Pre Specified Outcome: Serum Biomarkers of Sufficiency of Fat-soluble Vitamins - Vitamin D
Description: Vitamin D sufficiency is measured by the serum level of 25-hydroxy vitamin D
Time Frame: 24 Months
Population: as for outcome 10
Arm/Group | Corticosteroids | Placebo
Number analyzed (Participants) | 0 | 0

13. Other Pre Specified Outcome: Serum Biomarkers of Sufficiency of Fat-soluble Vitamins - Vitamin A
Description: Vitamin A sufficiency is defined as the molar ratio of serum retinol/retinol binding protein
Time Frame: 24 months
Population: as for outcome 10
Arm/Group | Corticosteroids | Placebo
Number analyzed (Participants) | 0 | 0

14. Other Pre Specified Outcome: Serum Biomarkers of Sufficiency of Fat-soluble Vitamins - Vitamin D
Description: Vitamin D sufficiency is measured by the serum level of 25-hydroxy vitamin D
Time Frame: 12 Months
Population: as for outcome 10
Arm/Group | Corticosteroids | Placebo
Number analyzed (Participants) | 0 | 0

15. Other Pre Specified Outcome: Serum Biomarkers of Sufficiency of Fat-soluble Vitamins - Vitamin K
Description: Vitamin K sufficiency is measured by INR (international normalized ratio)
Time Frame: 12 Months
Population: as for outcome 10
Arm/Group | Corticosteroids | Placebo
Number analyzed (Participants) | 0 | 0

16. Other Pre Specified Outcome: Serum Biomarkers of Sufficiency of Fat-soluble Vitamins - Vitamin E
Description: Vitamin E sufficiency is measured as the ratio of serum vitamin E/total lipids
Time Frame: 12 Months
Population: as for outcome 10
Arm/Group | Corticosteroids | Placebo
Number analyzed (Participants) | 0 | 0

17. Other Pre Specified Outcome: Serum Biomarkers of Sufficiency of Fat-soluble Vitamins - Vitamin A
Description: Vitamin A sufficiency is measured by the molar ratio of serum retinol/retinol binding protein
Time Frame: 12 months
Population: as for outcome 10
Arm/Group | Corticosteroids | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 24 months of age
Arm/Group | Corticosteroids | Placebo
Serious Adverse Events (participants affected / at risk) | 57/70 | 56/70
Other Adverse Events (participants affected / at risk) | 0/70 | 0/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Corticosteroids (N=70) | Placebo (N=70)
Congenital (Congenital, familial and genetic disorders) | 1 (1) | 1 (1) — AEs reported with regard to affected organ system
Gastrointestinal (Gastrointestinal disorders) | 5 (6) | 3 (3) — AEs reported with regard to affected organ system
Hepatic (Hepatobiliary disorders) | 22 (41) | 16 (30) — AEs reported with regard to affected organ system
Immunological (Immune system disorders) | 1 (1) | 0 (0) — AEs reported with regard to affected organ system
Infectious (Infections and infestations) | 50 (129) | 46 (109) — AEs reported with regard to affected organ system
Metabolic (Metabolism and nutrition disorders) | 1 (1) | 1 (2) — AEs reported as Metabolic
Miscellaneous (General disorders) | 3 (5) | 1 (1) — AEs reported with regard to affected organ system
Neoplastic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — AEs reported with regard to affected organ system
Neurological (Nervous system disorders) | 1 (1) | 0 (0) — AEs reported with regard to affected organ system
Nutritional (Metabolism and nutrition disorders) | 7 (8) | 9 (11) — AEs reported as Nutritional
Orthopedic (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) — AEs reported with regard to affected organ system
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — AEs reported with regard to affected organ system
Surgical (Surgical and medical procedures) | 7 (8) | 2 (2) — AEs reported with regard to affected organ system

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other